CLINICAL TRIAL: NCT01838863
Title: A Prospective, Randomized Comparison of Fresh Frozen Plasma Versus Standard Crystalloid Intravenous Fluid as Initial Resuscitation Fluid
Brief Title: Control of Major Bleeding After Trauma Study
Acronym: COMBAT
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Futility
Sponsor: Denver Health and Hospital Authority (Other)
Collaborators: U.S. Army Medical Research and Development Command (U.S. Federal Agency); University of Colorado, Denver (Other)
Responsible Party: Principal Investigator, Ernest E. Moore, MD, Professor and Vice Chair, Department of Surgery, Denver Health and Hospital Authority
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COMIRB# 12-1349; W81XWH1220028 (Other Grant/Funding Number: Department of Defense TATRC)
Record Dates: First submitted 2013-04-22; First posted 2013-04-24 (Estimated); Results first posted 2018-07-18 (Actual); Last update posted 2019-01-08 (Actual); Status verified 2018-12

CONDITIONS: Trauma; Hemorrhagic Shock
Keywords: coagulopathy; hemorrhagic shock; plasma; blood product transfusion
MeSH Terms: conditions — Wounds and Injuries; Shock, Hemorrhagic; Hemostatic Disorders | interventions — Standard of Care; Resuscitation; Saline Solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Plasma (Experimental): If the patient is randomized to experimental arm, 2 units of frozen type AB plasma (FP24) will be thawed in the Plasmatherm Dry Thawing and Warming Device according to the operator manual as approved by the FDA in the ambulance and infusion will commence as soon as the type AB plasma is ready, and will continue during transport to the emergency department (ED). After infusion of 2 units of type AB plasma is completed, subsequent care will proceed per institutional, Advanced Trauma Life Support (ATLS) guided resuscitation with acute packed red blood cells (pRBC) administration determined by the hemodynamic response and additional blood component administration guided by rapid thrombelastography (rTEG) and coagulation panel assessment in conjunction with clinical scenario.
  Interventions: Biological: Type AB plasma
- Standard (Active Comparator): If the patient is randomized to the standard arm, the patient will be given intravenous crystalloid fluid (normal saline) as the initial resuscitation fluid with 2 large bore IVs based on the current ATLS guidelines, the standard of care. Subsequent care will proceed per institutional, ATLS guided resuscitation with acute packed red blood cells pRBC administration determined by the hemodynamic response and additional blood component administration guided by rTEG and coagulation panel assessment in conjunction with clinical scenario.
  Interventions: Drug: Crystalloid fluid (standard of care for resuscitation)

INTERVENTIONS:
Biological: Type AB plasma — The plasma is thawed and administered to subjects in the experimental (plasma) arm.
  Other Names: Plasma frozen within 24 hours (FP24, PF24)
  Arms: Plasma
Drug: Crystalloid fluid (standard of care for resuscitation) — Normal saline will be give to subjects in the standard arm as the current standard of care for an initial resuscitation fluid
  Other Names: Normal saline
  Arms: Standard

SUMMARY:
Bleeding is the most avoidable cause of death in trauma patients. Up to one-third of severely injured trauma patients are found to be coagulopathic and forty percent of the mortality following severe injury is due to uncontrollable hemorrhage in the setting of coagulopathy. It has been established that early administration of fresh frozen plasma decreases mortality following severe injury, replacing lost coagulation factors, improving the coagulopathy and restoring blood volume. This study will determine if giving plasma to severely injured trauma patients during ambulance transport versus after arrival to the hospital will help reduce hemorrhage, thus decreasing both total blood product administration and mortality.

DETAILED DESCRIPTION:
Study Design: Severely injured trauma patients with a systolic blood pressure (SBP) ≤ 70 or SBP ≤ 90 with a heart rate ≥ 108 bpm at the scene will be enrolled and randomized to receive either 2 units of frozen plasma thawed in the field or normal saline (the current standard of care), as the initial resuscitation fluid. After this initial resuscitation fluid, both groups will receive the same standard of care, including packed red blood cells, additional normal saline, or plasma as needed based on laboratory and clinical evidence of coagulopathy. Blood samples and clinical information will be collected throughout the hospital stay up to 28 days after injury.

ELIGIBILITY:
Inclusion Criteria:

* Age>=18 years
* Acutely injured
* SBP<70 mmHg or SBP 71-90 mmHg with heart rate (HR)>108 beats per minute.

Exclusion Criteria:

* Visibly or verbally reported pregnant women
* known prisoners
* unsalvageable injuries (defined as asystolic or cardiopulmonary resuscitation prior to randomization)
* known objection to blood products
* the patient has an opt-out bracelet or, necklace or wallet card
* a family member present at the scene objects to the patient's enrollment in research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2014-04-07 (Actual); Primary Completion 2017-04-03 (Actual); Study Completion 2017-04-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ernest E Moore, MD, Principal Investigator — Denver Health Medical Center
Locations (1):
- Denver Health Medical Center, Denver, Colorado, United States

REFERENCES:
- [Derived] DeBot M, Erickson C, Schaid T, LaCroix I, Moore EE, Silliman C, Cohen MJ, D'Alessandro A, Hansen KC. Trauma-induced dysfibrinogenemia: the von Clauss assay does not accurately measure fibrinogen levels after injury. Blood Vessel Thromb Hemost. 2024 Jul 16;1(3):100017. doi: 10.1016/j.bvth.2024.100017. eCollection 2024 Sep. PMID 40766812
- [Derived] Pusateri AE, Moore EE, Moore HB, Le TD, Guyette FX, Chapman MP, Sauaia A, Ghasabyan A, Chandler J, McVaney K, Brown JB, Daley BJ, Miller RS, Harbrecht BG, Claridge JA, Phelan HA, Witham WR, Putnam AT, Sperry JL. Association of Prehospital Plasma Transfusion With Survival in Trauma Patients With Hemorrhagic Shock When Transport Times Are Longer Than 20 Minutes: A Post Hoc Analysis of the PAMPer and COMBAT Clinical Trials. JAMA Surg. 2020 Feb 1;155(2):e195085. doi: 10.1001/jamasurg.2019.5085. Epub 2020 Feb 19. PMID 31851290
- [Derived] Moore HB, Moore EE, Chapman MP, McVaney K, Bryskiewicz G, Blechar R, Chin T, Burlew CC, Pieracci F, West FB, Fleming CD, Ghasabyan A, Chandler J, Silliman CC, Banerjee A, Sauaia A. Plasma-first resuscitation to treat haemorrhagic shock during emergency ground transportation in an urban area: a randomised trial. Lancet. 2018 Jul 28;392(10144):283-291. doi: 10.1016/S0140-6736(18)31553-8. Epub 2018 Jul 20. PMID 30032977
- [Derived] Reynolds PS, Michael MJ, Cochran ED, Wegelin JA, Spiess BD. Prehospital use of plasma in traumatic hemorrhage (The PUPTH Trial): study protocol for a randomised controlled trial. Trials. 2015 Jul 30;16:321. doi: 10.1186/s13063-015-0844-5. PMID 26220293
- [Derived] Chapman MP, Moore EE, Chin TL, Ghasabyan A, Chandler J, Stringham J, Gonzalez E, Moore HB, Banerjee A, Silliman CC, Sauaia A. Combat: Initial Experience with a Randomized Clinical Trial of Plasma-Based Resuscitation in the Field for Traumatic Hemorrhagic Shock. Shock. 2015 Aug;44 Suppl 1(0 1):63-70. doi: 10.1097/SHK.0000000000000376. PMID 25784527

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The enrollment and randomization occurred almost simultaneously. Once the paramedics determined the patient to be eligible, the cooler was opened and the randomization was done based on the cooler content: cooler with plasma randomized the patient to the experimental and cooler with frozen water randomized the patient to the control group.
Groups:
- Plasma: If the patient is randomized to experimental arm, 2 units of frozen Type AB plasma (FP24) will be thawed in the Plasmatherm Dry Thawing and Warming Device according to the operator manual as approved by the FDA in the ambulance and infusion will commence as soon as the Type AB plasma is ready, and will continue during transport to the ED. After infusion of 2 units of Type AB plasma is completed, subsequent care will proceed per institutional, Advanced Trauma Life Support (ATLS) guided resuscitation with acute packed red blood cells (pRBC) administration determined by hemodynamic response and additional blood component administration guided by rapid thrombelastography (rTEG) and coagulation panel assessment in conjunction with clinical scenario.
  Type AB plasma: The plasma is thawed and administered to subjects in the experimental (plasma) arm.
- Standard: If the patient is randomized to the standard arm, the patient will be given intravenous crystalloid fluid (normal saline) as the initial resuscitation fluid with 2 large bore IVs based on the current ATLS guidelines, the standard of care. Subsequent care will proceed per institutional, ATLS guided resuscitation with acute pRBC administration determined by hemodynamic response and additional blood component administration guided by rTEG and coagulation panel assessment in conjunction with clinical scenario.
  Crystalloid fluid (standard of care for resuscitation): Normal saline will be give to subjects in the standard arm as the current standard of care for an initial resuscitation fluid
Period: Overall Study
Arm/Group | Plasma | Standard
Started | 75 | 69
Completed | 65 | 60
Not Completed | 10 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Plasma | Standard | Total
Number analyzed (Participants) | 65 | 60 | 125
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 33 [25 to 51] | 32.5 [25.8 to 42] | 33 [25 to 47]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 9 | 22
  Male | 52 | 51 | 103
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 34 | 39 | 73
  Not Hispanic or Latino | 31 | 21 | 52
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 65 | 60 | 125
Body Mass Index (BMI) [Median (Inter-Quartile Range); unit: kg/m^2] | 27.1 [23.9 to 30.5] | 26.1 [23.2 to 29.4] | 26.7 [23.4 to 30.5]
Comorbidities [Count of Participants; unit: Participants] — Presence of one or more additional diseases or disorders co-occurring in trauma patient.
  Participants | 10 | 8 | 18
Blunt injury mechanism [Count of Participants; unit: Participants] — Blunt force trauma is an injury that occurs when an object hits or strikes a part of the body.
  Participants | 30 | 32 | 62
New Injury Severity Scale (NISS) [Median (Inter-Quartile Range); unit: units on a scale] — The New Injury Severity Score (NISS) is an anatomical scoring system that provides an overall score for patients with multiple injuries. This is calculated as the sum of the squares of the top three Abbreviated Injury Scores (AIS) regardless of body region. AIS is an anatomical-based coding system on a scale of one to six, one being a minor injury and six being maximal. The NISS score takes values from 0 to 75. This score is virtually the only anatomical scoring system in use and correlates linearly with mortality, morbidity, hospital stay and other measures of severity.
  units on a scale | 27 [10 to 41] | 27 [11.8 to 35] | 27 [10 to 38]
Maximal Abbreviated Injury Score (AIS) for head and neck [Median (Inter-Quartile Range); unit: units on a scale] — Abbreviated Injury Score is an anatomical-based coding system on a scale of one to six, one being a minor injury and six being maximal.
  units on a scale | 0 [0 to 2] | 0 [0 to 2.3] | 0 [0 to 2]
Traumatic Brain Injury (TBI) defined as AIS head >=3 [Count of Participants; unit: Participants] | 15 | 13 | 28
Maximal Abbreviated Injury Score (AIS) chest [Median (Inter-Quartile Range); unit: units on a scale] — Abbreviated Injury Score is an anatomical-based coding system on a scale of one to six, one being a minor injury and six being maximal.
  units on a scale | 1 [0 to 3] | 3 [0 to 3] | 2 [0 to 3]
Maximal Abbreviated Injury Score (AIS) abdomen and pelvis [Median (Inter-Quartile Range); unit: units on a scale] — Abbreviated Injury Score is an anatomical-based coding system on a scale of one to six, one being a minor injury and six being maximal.
  units on a scale | 0 [0 to 3] | 0 [0 to 3] | 0 [0 to 3]
Maximal Abbreviated Injury Score (AIS) extremities [Median (Inter-Quartile Range); unit: units on a scale] — Abbreviated Injury Score is an anatomical-based coding system on a scale of one to six, one being a minor injury and six being maximal.
  units on a scale | 1 [0 to 3] | 0 [0 to 2] | 0 [0 to 2]
Heart rate (HR) in the field [Median (Inter-Quartile Range); unit: beats per minute (BPM)] | 110 [98 to 120] | 112 [100 to 120] | 110 [100 to 120]
Systolic blood pressure (SBP) in the field [Median (Inter-Quartile Range); unit: mmHg] | 64 [50 to 80] | 70 [58 to 80] | 68 [50 to 80]
Severe shock defined as systolic blood pressure (SBP) in the field <=70mmHg [Count of Participants; unit: Participants] | 44 | 33 | 77
Body temperature in the field [Median (Inter-Quartile Range); unit: degrees Celsius] — Population: The body temperature was measured in the field with a temporal scanner infrared thermometer. Due to the specifics of the study (acute trauma setting), it was not always possible to obtain a body temperature reading in the field (accident scene).
  degrees Celsius
    number analyzed (Participants) | 38 | 29 | 67
    (all) | 36 [34.8 to 36.6] | 36 [35.1 to 37] | 36 [34.9 to 36.9]
Glasgow Coma Scale (GCS) in the field [Median (Inter-Quartile Range); unit: units on a scale] — Glasgow Coma Scale (GCS) is a neurological scale which aims to give a reliable and objective way of recording the conscious state of a person for initial as well as subsequent assessment. The GCS is the summation of scores for eye, verbal, and motor responses. The minimum score is a 3 which indicates deep coma or a brain-dead state. The maximum is 15 which indicates a fully awake patient.
  units on a scale | 14 [7 to 15] | 14 [8 to 15] | 14 [8 to 15]
Haemoglobin (Hb) in the field [Median (Inter-Quartile Range); unit: g/dL] — Population: Due to the specifics of the study (acute trauma setting) it was not always possible to obtain a blood sample in the field (accident scene).
  g/dL
    number analyzed (Participants) | 32 | 27 | 59
    (all) | 15.1 [13.6 to 15.7] | 14.2 [13.2 to 15.9] | 14.6 [13.2 to 15.7]
Platelet count in the field [Median (Inter-Quartile Range); unit: 1000 cells/microL] — Population: Due to the specifics of the study (acute trauma setting) it was not always possible to obtain a blood sample in the field (accident scene).
  1000 cells/microL
    number analyzed (Participants) | 26 | 20 | 46
    (all) | 300.5 [251.8 to 353.2] | 273.5 [219 to 331] | 287.5 [245.5 to 345.8]
Fibrinogen in the field [Median (Inter-Quartile Range); unit: mg/dL] — Population: Due to the specifics of the study (acute trauma setting) it was not always possible to obtain a blood sample in the field (accident scene).
  mg/dL
    number analyzed (Participants) | 35 | 29 | 64
    (all) | 253 [226 to 308] | 278 [250 to 331] | 268 [228.5 to 322.5]
International normalized ratio (INR) in the field [Median (Inter-Quartile Range); unit: ratio] — Population: Measure Analysis Population Description: Defined as the first international normalized ratio (INR) obtained upon ED arrival. The international normalized ratio (INR) is an international standard for the prothrombin time (PT). This measures the time it takes for blood to clot. The normal range for a healthy person is 0.83-1.19.
  ratio
    number analyzed (Participants) | 36 | 29 | 65
    (all) | 1.1 [1 to 1.2] | 1.1 [1 to 1.1] | 1.1 [1 to 1.2]
International normalized ratio (INR) in the field >=1.3 [Count of Participants; unit: Participants] — Population: Due to the specifics of the study (acute trauma setting) it was not always possible to obtain a blood sample in the field (accident scene).
  Participants
    number analyzed (Participants) | 36 | 29 | 65
    (all) | 2 | 2 | 4
Partial thromboplastin time (PTT) in the field [Median (Inter-Quartile Range); unit: seconds] — Population: Due to the specifics of the study (acute trauma setting) it was not always possible to obtain a blood sample in the field (accident scene).
  seconds
    number analyzed (Participants) | 36 | 28 | 64
    (all) | 27.1 [25 to 30] | 26.9 [24.6 to 30.4] | 27.1 [24.7 to 30.4]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants That Died Within 28 Days Post Injury
Description: death within 28 days post injury (death of any cause except for death due to a second, clearly unrelated traumatic injury suffered after discharge)
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Plasma | Standard
Number analyzed (Participants) | 65 | 60
Participants | 10 | 6

2. Secondary Outcome: Composite Outcome of 28-day In-hospital Mortality and Postinjury Multiple Organ Failure (MOF) Incidence
Description: The occurrence of in-hospital death or MOF within the first 28 days postinjury. MOF is defined using the validated Denver MOF score (Denver MOF score>3 of simultaneously obtained scores after 48 hours postinjury).
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Plasma | Standard
Number analyzed (Participants) | 65 | 60
Participants | 14 | 7

3. Secondary Outcome: Admission Coagulopathy
Description: Defined as the first international normalized ratio (INR) obtained upon ED arrival. The international normalized ratio (INR) is an international standard for the prothrombin time (PT). This measures the time it takes for blood to clot. The normal range for a healthy person is 0.83-1.19. Usually, a high INR indicates a higher risk of bleeding, while a low INR suggests a higher risk of developing a clot.
Time Frame: within 30 minutes of Emergency Department (ED) arrival
Measure: Median (Inter-Quartile Range); unit: ratio
Arm/Group | Plasma | Standard
Number analyzed (Participants) | 63 | 58
ratio | 1.27 [1.11 to 1.4] | 1.15 [1.08 to 1.29]

4. Secondary Outcome: Number of Participants With Admission Severe Coagulopathy
Description: Defined as international normalized ratio (INR) >1.3 obtained upon ED arrival. The international normalized ratio (INR) is an international standard for the prothrombin time (PT). This measures the time it takes for blood to clot. The normal range for a healthy person is 0.83-1.19. Usually, a high INR indicates a higher risk of bleeding, while a low INR suggests a higher risk of developing a clot.
Time Frame: within 30 minutes of Emergency Department (ED) arrival
Measure: Count of Participants; unit: Participants
Arm/Group | Plasma | Standard
Number analyzed (Participants) | 63 | 58
Participants | 28 | 14

5. Secondary Outcome: Admission Clot Strength
Description: Admission clot strength will be measured by thrombelastography G-value upon ED arrival. Clot strength measured in kilodynes per square centimetre (kdyn/cm^2).
Time Frame: within 30 minutes of ED arrival
Measure: Median (Inter-Quartile Range); unit: kdyne/cm^2
Arm/Group | Plasma | Standard
Number analyzed (Participants) | 55 | 51
kdyne/cm^2 | 7.7 [6.2 to 8.9] | 7.1 [5.4 to 9.7]

6. Secondary Outcome: Admission Acidosis
Description: Admission acidosis measured by lactate upon ED arrival.
Time Frame: within 30 minutes of ED arrival
Measure: Median (Inter-Quartile Range); unit: mmol/L
Arm/Group | Plasma | Standard
Number analyzed (Participants) | 53 | 52
mmol/L | 5.5 [3.9 to 8.5] | 4.9 [3.2 to 7]

7. Secondary Outcome: Number of Participants With Admission Severe Acidosis
Description: Admission severe acidosis measured by lactate>5 upon ED arrival.
Time Frame: within 30 minutes of ED arrival
Measure: Count of Participants; unit: Participants
Arm/Group | Plasma | Standard
Number analyzed (Participants) | 53 | 52
Participants | 27 | 25

8. Secondary Outcome: Admission Acidosis
Description: Admission acidosis will be defined by base deficit (BD) upon ED arrival.
Time Frame: within 30 minutes of ED arrival
Measure: Median (Inter-Quartile Range); unit: mEq/L
Arm/Group | Plasma | Standard
Number analyzed (Participants) | 51 | 50
mEq/L | 9 [5.5 to 13] | 8.8 [6 to 13]

9. Secondary Outcome: Number of Participants With Admission Severe Acidosis
Description: Admission severe acidosis will be defined by base deficit (BD>10) upon ED arrival.
Time Frame: within 30 minutes of ED arrival
Measure: Count of Participants; unit: Participants
Arm/Group | Plasma | Standard
Number analyzed (Participants) | 51 | 50
Participants | 21 | 22

10. Other Pre Specified Outcome: Baseline (Field) Coagulation Factor Levels
Description: defined as the first coagulation factor level obtained in the field prior to intervention
  Coagulation Factor Reference Ranges
  F2 F5 F7 F8 F9 F11
  * % % % % % % 67.0 - 107.0 63.0 - 116.0 52.0 - 120.0 58.0 - 132.0 47.0 - 122.0 52.0 - 120.0
Time Frame: after injury and prior to hospital arrival, at about 15 minutes after injury
Measure: Median (Inter-Quartile Range); unit: percentage of activity
Arm/Group | Plasma | Standard
Number analyzed (Participants) | 34 | 26
percentage of activity
  Coagulation factor II (prothrombin) | 95 [85 to 105] | 98 [85 to 105]
  Coagulation factor V (proaccelerin) | 85 [73 to 99] | 91.5 [77 to 100]
  Coagulation factor VII (proconvertin) | 101.5 [84 to 127] | 89.5 [80 to 114]
  Coagulation factor VIII (antihemophilic factor) | 396.8 [273 to 476] | 411.8 [353.2 to 464.6]
  Coagulation factor IX (plasma thromboplastin comp) | 157 [128 to 180] | 160.5 [148 to 174]
  Coagulation factor XI (plasma thromboplastin ante) | 126.5 [106 to 153] | 141.5 [100 to 168]

11. Other Pre Specified Outcome: Number of Participants With Abnormal Baseline (Field) Coagulation Factor XIII Level
Description: defined as abnormal coagulation factor XIII level obtained in the field prior to intervention
Time Frame: after injury prior to hospital arrival
Measure: Count of Participants; unit: Participants
Arm/Group | Plasma | Standard
Number analyzed (Participants) | 34 | 26
Participants | 0 | 0

12. Other Pre Specified Outcome: Admission (First Arrival) Coagulation Factor Levels
Description: defined as the first coagulation factor level obtained upon ED arrival
  Coagulation Factor Reference Ranges
  F2 F5 F7 F8 F9 F11
  * % % % % % % 67.0 - 107.0 63.0 - 116.0 52.0 - 120.0 58.0 - 132.0 47.0 - 122.0 52.0 - 120.0
Time Frame: after injury prior to hospital arrival
Population: Not all the timepoints are available for all the patients.
Measure: Median (Inter-Quartile Range); unit: percentage of activity
Arm/Group | Plasma | Standard
Number analyzed (Participants) | 47 | 41
percentage of activity
  Coagulation factor I (fibrinogen): number analyzed (Participants) | 39 | 40
  Coagulation factor I (fibrinogen) | 195 [157 to 275] | 222 [154.5 to 282]
  Coagulation factor II (prothrombin) | 71 [57 to 88] | 79 [65 to 92]
  Coagulation factor V (proaccelerin) | 64 [41 to 83] | 69 [52 to 91]
  Coagulation factor VII (proconvertin) | 72 [56 to 94] | 74 [52 to 94]
  Coagulation factor VIII (antihemophilic factor) | 283.4 [168.4 to 434.2] | 355.2 [279 to 462.6]
  Coagulation factor IX (plasma thromboplastin comp) | 121 [87 to 142] | 135 [99 to 159]
  Coagulation factor XI (plasma thromboplastin ante) | 81 [58 to 127] | 109 [72 to 135]

13. Other Pre Specified Outcome: Number of Participants With Abnormal Admission Coagulation Factor XIII (Fibrin-stabilizing Factor) Level
Description: defined as the first abnormal factor XIII (fibrin-stabilizing factor) level obtained upon ED arrival
Time Frame: within 30 minutes of Emergency Department (ED) arrival
Measure: Count of Participants; unit: Participants
Arm/Group | Plasma | Standard
Number analyzed (Participants) | 39 | 40
Participants | 0 | 2

14. Other Pre Specified Outcome: Exploratory Analyses
Description: Number of participants with 24-hour mortality, adverse outcome free days and transfusions
Time Frame: Hospital stay up to 28 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Plasma | Standard
Number analyzed (Participants) | 65 | 60
Participants
  24-hour mortality | 8 | 6
  Acute lung injury (ALI) within 28 days | 18 | 12
  Acute lung injury (ALI) within 6 hours post-transf | 19 | 22
  MOF (Denver MOF score>3) | 4 | 1
  Haemoglobin (Hb)<7g/dL within 6 hours | 3 | 2
  Required red blood cell transf. within 24 hour | 36 | 35
  Massive transf. (>=10 units of RBC or death/6 hrs | 15 | 12
  Required plasma in first 24 h (not counting field) | 29 | 26
  Required platelets in first 24 h | 15 | 11
  Required cryoprecipitate in first 24 h | 8 | 4
  Required tranexamic acid (TXA) in first 6 h | 6 | 7
  Required factor VII infusion in first 24 h | 1 | 0

15. Other Pre Specified Outcome: Exploratory Analyses.
Description: Adverse outcome free days
Time Frame: Hospital stay up to 28 days.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Plasma | Standard
Number analyzed (Participants) | 65 | 60
days
  Ventilator free days | 26 [11 to 28] | 26 [18 to 28]
  Intensive care unit (ICU) free days | 23 [7 to 26] | 24 [16.5 to 26]

16. Other Pre Specified Outcome: Number of Participants With Mortality, Adverse Outcome-free Days and Transfusions in the Sub-group With Less Severe Hemorrhagic Shock
Description: Mortality, adverse outcome-free days and transfusions in the patients with initial systolic blood pressure (SBP) 71-90 mmHg and heart rate (HR) of 108 or greater
Time Frame: Hospital stay up to 28 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Plasma | Standard
Number analyzed (Participants) | 21 | 27
Participants
  28-day mortality | 0 | 2
  Death or multiple organ failure within 28 days | 0 | 2
  Acute lung injury (ALI) within 28 days | 8 | 12
  Acute lung injury (ALI) within 6 h post-transfusio | 5 | 8
  MOF (Denver MOF score>3) | 0 | 0
  Haemoglobin (Hb)<7g/dL within 6 hours | 1 | 0
  Required red blood cell transfusion within 24 h | 7 | 14
  Massive transf. (>=10 units of RBC or death/6 hrs | 0 | 5
  Required plasma in first 24 h (not counting field) | 3 | 9
  Required platelets in first 24 h | 1 | 6
  Required cryoprecipitate in first 24 h | 0 | 2
  Required tranexamic acid (TXA) in first 6 h | 2 | 2
  Required factor VII infusion in first 24 h | 0 | 0

17. Other Pre Specified Outcome: Adverse Outcome-free Days in a Sub-group With Less Severe Hemorrhagic Shock
Description: Adverse outcome-free days in the patients with initial systolic blood pressure (SBP) 71-90 mmHg and heart rate (HR) of 108 or greater
Time Frame: Hospital stay up to 28 days.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Plasma | Standard
Number analyzed (Participants) | 21 | 27
days
  Ventilator free days | 27 [22 to 28] | 26 [17 to 28]
  Intensive care unit (ICU) free days | 24 [22 to 27] | 25 [12 to 26]

18. Other Pre Specified Outcome: Level of Haemoglobin (Hb) in a Sub-group With Less Severe Hemorrhagic Shock
Description: Level of Haemoglobin (Hb) in g/dL in the patients with initial systolic blood pressure (SBP) 71-90 mmHg and heart rate (HR) of 108 or greater
Time Frame: Hospital stay up to 28 days.
Measure: Median (Inter-Quartile Range); unit: g/dL
Arm/Group | Plasma | Standard
Number analyzed (Participants) | 21 | 27
g/dL
  Admission (first arrival) Haemoglobin (Hb) | 14.4 [13 to 15.2] | 13.5 [12 to 14.7]
  Lowest Haemoglobin (Hb) in first 6 hours | 11.6 [10.1 to 13.6] | 11.4 [9.3 to 13]

19. Other Pre Specified Outcome: Blood Product Transfusion in a Sub-group With Less Severe Hemorrhagic Shock
Description: Transfusions of blood products in units in the patients with initial systolic blood pressure (SBP) 71-90 mmHg and heart rate (HR) of 108 or greater
Time Frame: Hospital stay up to 28 days.
Measure: Median (Inter-Quartile Range); unit: units
Arm/Group | Plasma | Standard
Number analyzed (Participants) | 21 | 27
units
  Red blood cell (RBC) transfusion in 24 h | 0 [0 to 2] | 1 [0 to 8]
  Plasma transfused in 24h (excluding pre-admission) | 0 [0 to 0] | 0 [0 to 2]
  Platelets transfused in 24 h | 0 [0 to 0] | 0 [0 to 0]
  Cryoprecipitate transfused in 24 h | 0 [0 to 0] | 0 [0 to 0]

20. Other Pre Specified Outcome: Time to Admission and First Blood Transfusion in a Sub-group With Less Severe Hemorrhagic Shock
Description: Time to Admission and First Blood Transfusion in minutes in the patients with initial systolic blood pressure (SBP) 71-90 mmHg and heart rate (HR) of 108 or greater
Time Frame: Hospital stay up to 28 days.
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Plasma | Standard
Number analyzed (Participants) | 21 | 27
minutes
  Time from injury to ED admission | 30 [25 to 40] | 25 [19 to 32]
  Time from injury to first unit of RBC | 119.5 [44.5 to 159.5] | 39 [24 to 56]

21. Other Pre Specified Outcome: Number of Participants With Mortality, Adverse Outcome-free Days and Transfusions in a Sub-group With Severe Hemorrhagic Shock
Description: Mortality, adverse outcome-free days and transfusions in the patients with initial systolic blood pressure (SBP) <=70 mmHg
Time Frame: Hospital stay up to 28 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Plasma | Standard
Number analyzed (Participants) | 44 | 33
Participants
  28-day mortality | 10 | 4
  Death or multiple organ failure within 28 days | 14 | 5
  24-hour mortality | 8 | 4
  Acute lung injury (ALI) within 28 days | 20 | 18
  Acute lung injury (ALI) within 6 h post-transfusio | 14 | 14
  MOF (Denver MOF score>3) | 4 | 1
  Haemoglobin (Hb)<7g/dL within 6 hours | 2 | 2
  Required red blood cell transfusion within 24 h | 29 | 21
  Massive transf. (>=10 units of RBC or death/6 hrs | 15 | 7
  Required plasma in first 24 h (not counting field) | 26 | 17
  Required platelets in first 24 h | 12 | 4
  Required cryoprecipitate in first 24 h | 8 | 2
  Required tranexamic acid (TXA) in first 6 h | 4 | 5
  Required factor VII infusion in first 24 h | 1 | 0

22. Other Pre Specified Outcome: Number of Adverse Outcome Free Days in a Sub-group With Severe Hemorrhagic Shock
Description: Adverse outcome-free days in the patients with initial systolic blood pressure (SBP) <=70 mmHg
Time Frame: Hospital stay up to 28 days.
Population: Not all the timepoints are available for all the patients.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Plasma | Standard
Number analyzed (Participants) | 44 | 33
days
  Ventilator free days | 24.5 [0 to 27.5] | 26 [22 to 28]
  Intensive care unit (ICU) free days | 20 [0 to 26] | 23 [19 to 25]

23. Other Pre Specified Outcome: Number of Participants in a Sub-group With no Severe Traumatic Brain Injury (TBI)
Description: Number of participants with mortality, adverse outcome-free days and transfusions in the patients with no severe traumatic brain injury (TBI) is defined as Abbreviated Injury Score (AIS) for Head/Neck >=3.
Time Frame: Hospital stay up to 28 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Plasma | Standard
Number analyzed (Participants) | 52 | 45
Participants
  28-day mortality | 6 | 5
  Death or multiple organ failure within 28 days | 9 | 6
  24-hour mortality | 6 | 5
  Acute lung injury (ALI) within 28 days | 20 | 21
  Possible transfusion associated acute lung injury | 12 | 16
  Required red blood cell transfusion within 72 h | 28 | 26
  Massive transf. (>=10 units of RBC or death/6 hrs | 10 | 10
  Required tranexamic acid (TXA) in first 6 h | 5 | 6
  Required factor VII infusion in first 24 h | 1 | 0

24. Other Pre Specified Outcome: Exploratory Analyses in a Sub-group With Severe Traumatic Brain Injury (TBI)
Description: Number of participants with 28-day mortality. Traumatic brain injury (TBI) is defined as Abbreviated Injury Score (AIS) for Head/Neck >=3.
Time Frame: Hospital stay up to 28 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Plasma | Standard
Number analyzed (Participants) | 13 | 15
Participants | 4 | 1

25. Other Pre Specified Outcome: Severe Adverse Events (SAE)
Description: Number of participants with severe adverse events (SAE)
Time Frame: Hospital stay up to day 28
Measure: Count of Participants; unit: Participants
Arm/Group | Plasma | Standard
Number analyzed (Participants) | 75 | 69
Participants
  Any SAEs | 34 | 24
  Death | 12 | 6
  Infections | 14 | 13
  Thromboembolic events | 4 | 2
  Non-infectious and non-thromboembolic events | 15 | 11
  MOF (Denver MOF score>3) | 5 | 1
  Organ failure (not MOF) | 15 | 13

26. Other Pre Specified Outcome: Haemoglobin (Hb) Level in a Sub-group With Severe Hemorrhagic Shock
Description: Haemoglobin (Hb) level in the patients with initial systolic blood pressure (SBP) <=70 mmHg
Time Frame: Hospital stay up to 28 days.
Population: Not all the timepoints are available for all the patients.
Measure: Median (Inter-Quartile Range); unit: g/dL
Arm/Group | Plasma | Standard
Number analyzed (Participants) | 44 | 33
g/dL
  Admission (first arrival) Haemoglobin (Hb) | 11.8 [10.5 to 13.8] | 13.2 [11.8 to 14.6]
  Lowest Haemoglobin (Hb) in first 6 hours | 11.3 [8.7 to 12.4] | 10.8 [8.7 to 12.5]

27. Other Pre Specified Outcome: Blood Product Transfusion in a Sub-group With Severe Hemorrhagic Shock
Description: Number of blood products transfused in units in the patients with initial systolic blood pressure (SBP) <=70 mmHg
Time Frame: Hospital stay up to 28 days.
Population: Not all the timepoints are available for all the patients.
Measure: Median (Inter-Quartile Range); unit: units
Arm/Group | Plasma | Standard
Number analyzed (Participants) | 44 | 33
units
  Red blood cell (RBC) transfusion in 24 h | 3.5 [0 to 13.5] | 3 [0 to 8]
  Plasma transfused in 24h (excluding pre-admission) | 1 [0 to 5] | 1 [0 to 3]
  Platelets transfused in 24 h | 0 [0 to 1] | 0 [0 to 0]
  Cryoprecipitate transfused in 24 h | 0 [0 to 0] | 0 [0 to 0]

28. Other Pre Specified Outcome: Time to Admission and First Blood Transfusion in a Sub-group With Severe Hemorrhagic Shock
Description: Time to Admission and First Blood Transfusion in the patients with initial systolic blood pressure (SBP) <=70 mmHg
Time Frame: Hospital stay up to 28 days.
Population: Not all the timepoints are available for all the patients.
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Plasma | Standard
Number analyzed (Participants) | 44 | 33
minutes
  Time from injury to ED admission | 28 [21 to 33] | 23 [19 to 28]
  Time from injury to first unit of RBC | 48 [32 to 59] | 36 [30 to 44]

29. Other Pre Specified Outcome: Haemoglobin (Hb) Level
Description: Haemoglobin (Hb) level in g/dL units.
Time Frame: Hospital stay up to 28 days.
Measure: Median (Inter-Quartile Range); unit: g/dL
Arm/Group | Plasma | Standard
Number analyzed (Participants) | 65 | 60
g/dL
  Admission (first arrival) Haemoglobin (Hb) | 12.6 [11.3 to 14.7] | 13.5 [11.9 to 14.7]
  Lowest Haemoglobin (Hb) in first 6 hours | 11.3 [9.6 to 12.6] | 11 [9.1 to 12.8]

30. Other Pre Specified Outcome: Number of Blood Products Transfused.
Description: Number of blood products transfused in units.
Time Frame: Hospital stay up to 28 days.
Measure: Median (Inter-Quartile Range); unit: units
Arm/Group | Plasma | Standard
Number analyzed (Participants) | 65 | 60
units
  Red blood cell (RBC) transfusion in 24 h | 2 [0 to 8] | 1.5 [0 to 8]
  Plasma transfused in 24h (excluding pre-admission) | 0 [0 to 4] | 0 [0 to 3]
  Platelets transfused in 24 h | 0 [0 to 0] | 0 [0 to 0]
  Cryoprecipitate transfused in 24 h | 0 [0 to 0] | 0 [0 to 0]

31. Other Pre Specified Outcome: Time to Admission and First Blood Transfusion
Description: Time to admission and first blood product transfusion in minutes.
Time Frame: Hospital stay up to 28 days.
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Plasma | Standard
Number analyzed (Participants) | 65 | 60
minutes
  Time from injury to ED admission | 28 [22 to 34] | 24 [19 to 31]
  Time from injury to first unit of RBC | 46.5 [32 to 55.5] | 37 [24 to 46]
  Time from ED admission to first unit of RBC | 16 [7 to 28] | 10 [4 to 18]
  Time to first plasma (including pre-admission) | 24 [20 to 31.5] | 58.5 [40 to 115]
  Time from admission to first platelet transfused | 130 [91 to 222] | 88 [56 to 166]

32. Post Hoc Outcome: Baseline (Field) Citrated Rapid Thrombelastography (CR-TEG) Parameters.
Description: Baseline (field) sample drawn prior to intervention in the field and measured by citrated rapid thrombelastography (CR-TEG) activated clotting time (ACT).
Time Frame: after injury and prior to hospital arrival, at about 15 minutes after injury
Measure: Median (Inter-Quartile Range); unit: second
Arm/Group | Plasma | Standard
Number analyzed (Participants) | 43 | 37
second | 121 [113 to 128] | 121 [113 to 128]

33. Post Hoc Outcome: Admission (ED) Citrated Rapid Thrombelastography (CR-TEG) Parameters.
Description: Admission (ED) sample drawn upon ED admission and measured by citrated rapid thrombelastography (CR-TEG) activated clotting time (ACT) in seconds.
Time Frame: post-intervention and upon ED arrival
Measure: Median (Inter-Quartile Range); unit: second
Arm/Group | Plasma | Standard
Number analyzed (Participants) | 55 | 51
second | 128 [113 to 136] | 121 [113 to 136]

34. Post Hoc Outcome: Baseline (Field) Citrated Rapid Thrombelastography (CR-TEG) Parameters.
Description: Baseline (field) sample drawn prior to intervention in the field and measured by citrated rapid thrombelastography (CR-TEG) angle in degrees.
Time Frame: after injury and prior to hospital arrival, at about 15 minutes after injury
Measure: Median (Inter-Quartile Range); unit: degrees
Arm/Group | Plasma | Standard
Number analyzed (Participants) | 43 | 37
degrees | 70.6 [66.9 to 75.6] | 70.6 [66.1 to 74.3]

35. Post Hoc Outcome: Baseline (Field) Citrated Rapid Thrombelastography (CR-TEG) Parameters.
Description: Baseline (field) sample drawn prior to intervention in the field and measured by citrated rapid thrombelastography (CR-TEG) maximum amplitude (MA).
Time Frame: after injury and prior to hospital arrival, at about 15 minutes after injury
Measure: Median (Inter-Quartile Range); unit: millimeter (mm)
Arm/Group | Plasma | Standard
Number analyzed (Participants) | 43 | 37
millimeter (mm) | 62 [57.5 to 68] | 63.5 [58 to 67]

36. Post Hoc Outcome: Baseline (Field) Citrated Rapid Thrombelastography (CR-TEG) Parameters.
Description: Baseline (field) sample drawn prior to intervention in the field and measured by citrated rapid thrombelastography (CR-TEG). Clot strength measured in kilodynes per square centimetre (kdyn/cm^2).
Time Frame: after injury and prior to hospital arrival, at about 15 minutes after injury
Measure: Median (Inter-Quartile Range); unit: kdyn/cm^2
Arm/Group | Plasma | Standard
Number analyzed (Participants) | 43 | 37
kdyn/cm^2 | 8.2 [6.8 to 10.6] | 8.7 [6.9 to 10.2]

37. Post Hoc Outcome: Baseline (Field) Citrated Rapid Thrombelastography (CR-TEG) Parameters.
Description: Baseline (field) sample drawn prior to intervention in the field and measured by citrated rapid thrombelastography (CR-TEG). Percentage of clot lysis 30 minutes after maximal amplitude (MA) value is finalized.
Time Frame: after injury and prior to hospital arrival, at about 15 minutes after injury
Measure: Median (Inter-Quartile Range); unit: percentage of clot lysed at 30 minutes
Arm/Group | Plasma | Standard
Number analyzed (Participants) | 43 | 37
percentage of clot lysed at 30 minutes | 2.2 [1 to 3.7] | 1.8 [0.9 to 3.7]

38. Post Hoc Outcome: Admission (ED) Citrated Rapid Thrombelastography (CR-TEG) Parameters.
Description: Admission (ED) sample drawn upon ED admission and measured by citrated rapid thrombelastography (CR-TEG) angle measured in degrees.
Time Frame: post-intervention and upon ED arrival
Measure: Median (Inter-Quartile Range); unit: degree
Arm/Group | Plasma | Standard
Number analyzed (Participants) | 55 | 51
degree | 60.5 [55.5 to 64] | 58.5 [52 to 66]

39. Post Hoc Outcome: Admission (ED) Citrated Rapid Thrombelastography (CR-TEG) Parameters.
Description: Admission (ED) sample drawn upon ED admission and measured by citrated rapid thrombelastography (CR-TEG) maximal amplitude (MA).
Time Frame: post-intervention and upon ED arrival
Measure: Median (Inter-Quartile Range); unit: millimeter (mm)
Arm/Group | Plasma | Standard
Number analyzed (Participants) | 55 | 51
millimeter (mm) | 70.9 [66.1 to 76.1] | 69.3 [63.2 to 74.4]

40. Post Hoc Outcome: Admission (ED) Citrated Rapid Thrombelastography (CR-TEG) Parameters.
Description: Admission (ED) sample drawn upon ED admission and measured by citrated rapid thrombelastography (CR-TEG) clot strength measures by G value in kilodynes per square centimetre (kdyn/cm^2).
Time Frame: post-intervention and upon ED arrival
Measure: Median (Inter-Quartile Range); unit: kdyn/cm^2
Arm/Group | Plasma | Standard
Number analyzed (Participants) | 55 | 51
kdyn/cm^2 | 7.7 [6.2 to 8.9] | 7.1 [5.4 to 9.7]

41. Post Hoc Outcome: Admission (ED) Citrated Rapid Thrombelastography (CR-TEG) Parameters.
Description: Admission (ED) sample drawn upon ED admission and measured by citrated rapid thrombelastography (CR-TEG) clot lysis 30 minutes after the maximal amplitude (MA) was finalized.
Time Frame: post-intervention and upon ED arrival
Measure: Median (Inter-Quartile Range); unit: percentage of clot lysed at 30 minutes
Arm/Group | Plasma | Standard
Number analyzed (Participants) | 55 | 51
percentage of clot lysed at 30 minutes | 1.3 [0.3 to 2.6] | 1.6 [0.7 to 3.1]

ADVERSE EVENTS:
Time Frame: Hospital stay up to 28 days.
Arm/Group | Plasma | Standard
All-Cause Mortality (participants affected / at risk) | 12/75 | 6/69
Serious Adverse Events (participants affected / at risk) | 34/75 | 24/69
Other Adverse Events (participants affected / at risk) | 5/75 | 2/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Plasma (N=75) | Standard (N=69)
Infections (Infections and infestations) | 14 (23) | 13 (20)
DVTs and PEs (Vascular disorders) | 4 (4) | 2 (2) — Deep venous thrombosis (DVT), pulmonary embolism (PE) and pulmonary infarction (PI).
Acute kidney injury (AKI) (Renal and urinary disorders) | 5 (5) | 6 (6) — Acute kidney injury (AKI), kidney failure and renal artery pseudoaneurysm.
Acute respiratory distress syndrome (ARDS) (Respiratory, thoracic and mediastinal disorders) | 20 (20) | 14 (14) — Acute respiratory distress syndrome (ARDS) and lung failure
Liver failure (Hepatobiliary disorders) | 4 (4) | 4 (4) — Liver failure and bile duct leak
Cardiac (Cardiac disorders) | 7 (7) | 6 (6) — Organ failure, atrial fibrillation and ventricular tachycardia
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0)
GI bleed (Gastrointestinal disorders) | 2 (2) | 0 (0) — Gastrointestinal bleeding and abdominal compartment syndrome
Hematoma (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Pre-sacral hematoma
Hemorrhage (Surgical and medical procedures) | 2 (2) | 0 (0) — Delayed hemorrhage from surgical site and torn suture
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Plasma (N=75) | Standard (N=69)
Intensive Care Unit (ICU) delirium (Psychiatric disorders) | 3 | 2
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0
Facial paralysis (Nervous system disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-12-27): https://cdn.clinicaltrials.gov/large-docs/63/NCT01838863/Prot_SAP_000.pdf
  • Informed Consent Form (2017-02-07): https://cdn.clinicaltrials.gov/large-docs/63/NCT01838863/ICF_001.pdf